CLINICAL TRIAL: NCT04528160
Title: Pain Neuroscience Education for Older Adults With Pain From Primary Care: a Feasibility Study
Brief Title: Pain Neuroscience Education for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, Anabela G Silva, Assistant Professor, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PNE4OlderAdults
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain neuroscience education and exercise (Experimental): This group will receive an 8-week intervention (1 session per week) of pain neuroscience education and exercise.
  PNE will be conducted in line with international guidelines and will cover the neurophysiology of pain, transition from acute to chronic pain and the nervous system ability to modulate the pain experience. Exercise will include mobility, balance and strength exercises.
  Interventions: Other: Pain neuroscience education and exercise
- Usual care (Active Comparator): This group will receive usual care administered by general practitioners at primary care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Pain neuroscience education and exercise — PNE will be conducted in line with international guidelines and will cover the neurophysiology of pain, transition from acute to chronic pain and the nervous system ability to modulate the pain experience. Exercise will included genera exercise delivered at moderate intensity.
  Arms: Pain neuroscience education and exercise
Other: Usual Care — Usual care delivered at primary care for older adults with pain.
  Arms: Usual care

SUMMARY:
This study aims to investigate the feasibility of using pain neuroscience education for older adults with chronic pain from primary care services. It will have a group of participants receiving pain neuroscience education and exercise and a group receiving usual care.

ELIGIBILITY:
Inclusion Criteria:

* be able to read and write and have chronic pain (defined as pain lasting 3 months or more and felt at least once a week during these 3 months ) anywhere in the body.

Exclusion Criteria:

* presence of pathology of the nervous or cardiovascular systems, cancer, or having had a surgery in the last 6 months or the presence of a condition for which the practice of therapeutic exercise could be contraindicated.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Inclusion rate | 9 weeks
  ratio between the number of participants included in the study and the total number of people contacted
Refusal rate | 9 weeks
  ratio between the number of individuals who refused to participate in the study and the number of individuals contacted
Exclusion rate | 9 weeks
  ratio between the number of individuals excluded for not meeting the inclusion criteria and the total number of individuals contacted
Dropout rate | 9 weeks
  ratio between the number of participants who abandoned the study and the number of participants who completed the initial assessment
Retention rate | 9 weeks
  ratio between the number of participants who completed the final assessment and the number of participants who completed the initial assessment
Number of participants reporting adverse events | 9 weeks
  Self-report of any adverse event perceived as being related to the intervention
Perception of participants towards the intervention structure and content | 9 weeks
  Semi-structured interviews with participants on the structure and content of the intervention

SECONDARY OUTCOMES:
Pain severity and interference | Baseline
  Assessed using the Brief Pain Inventory questionnaire (range 0-110 and higher values are indicative of higher pain severity and interference)
Pain severity and interference | 9 weeks
  Assessed using the Brief Pain Inventory questionnaire (range 0-110 and higher values are indicative of higher pain severity and interference)
Pain severity and interference | 6 months
  Assessed using the Brief Pain Inventory questionnaire (range 0-110 and higher values are indicative of higher pain severity and interference)
Pain catastrophizing | Baseline
  Assessed using the Pain Catastrophizing Scale (range 0-52 and higher values are indicative of higher pain catastrophizing)
Pain catastrophizing | 9 weeks
  Assessed using the Pain Catastrophizing Scale (range 0-52 and higher values are indicative of higher pain catastrophizing)
Pain catastrophizing | 6 months
  Assessed using the Pain Catastrophizing Scale (range 0-52 and higher values are indicative of higher pain catastrophizing)
Depression | Baseline
  Assessed using the Geriatric Depression Scale (range 0-15 and values of 5 or higher are indicative of depression)
Depression | 9 weeks
  Assessed using the Geriatric Depression Scale (range 0-15 and values of 5 or higher are indicative of depression)
Depression | 6 months
  Assessed using the Geriatric Depression Scale (range 0-15 and values of 5 or higher are indicative of depression)
Fear of movement | Baseline
  Assessed using the TAMPA Scale, which assesses fear of movement (range: 13-52 and higher values are indicative of higher levels of fear of movement)
Fear of movement | 6 weeks
  Assessed using the TAMPA Scale, which assesses fear of movement (range: 13-52 and higher values are indicative of higher levels of fear of movement)
Fear of movement | 6 months
  Assessed using the TAMPA Scale, which assesses fear of movement (range: 13-52 and higher values are indicative of higher levels of fear of movement)
Knowledge of pain neuroscience | Baseline
  Assessed using the pain neurophysiology questionnaire (range 0-19 and higher values are indicative of more knowledge on pain neurophysiology)
Knowledge of pain neuroscience | 9 weeks
  Assessed using the pain neurophysiology questionnaire (range 0-19 and higher values are indicative of more knowledge on pain neurophysiology)
Knowledge of pain neuroscience | 6 months
  Assessed using the pain neurophysiology questionnaire (range 0-19 and higher values are indicative of more knowledge on pain neurophysiology)
Gait velocity | Baseline
  Assessed using the gait velocity test - the time, in seconds, that each participant takes to walk 4 meters
Gait velocity | 9 weeks
  Assessed using the gait velocity test - the time, in seconds, that each participant takes to walk 4 meters
Gait velocity | 6 months
  Assessed using the gait velocity test - the time, in seconds, that each participant takes to walk 4 meters
Postural control | Baseline
  Assessed using the Timed up and go test - the time, in seconds, that it takes to stand from a chair, walk 3 meters, turn, walk another 3 meters to sit in the chair.
Postural control | 9 weeks
  Assessed using the Timed up and go test - the time, in seconds, that it takes to stand from a chair, walk 3 meters, turn, walk another 3 meters to sit in the chair.
Postural control | 6 months
  Assessed using the Timed up and go test - the time, in seconds, that it takes to stand from a chair, walk 3 meters, turn, walk another 3 meters to sit in the chair.
Self-perceived disability | Baseline
  assessed using the World Health Organization Disability Assessment Schedule 2.0 - 12-item version of WHODAS 2.0) questionnaire (range: 12-60 and higher values are indicative of higher levels of disability)
Self-perceived disability | 9 weeks
  assessed using the World Health Organization Disability Assessment Schedule 2.0 - 12-item version of WHODAS 2.0) questionnaire (range: 12-60 and higher values are indicative of higher levels of disability)
Self-perceived disability | 6 months
  assessed using the World Health Organization Disability Assessment Schedule 2.0 - 12-item version of WHODAS 2.0) questionnaire (range: 12-60 and higher values are indicative of higher levels of disability)
Perception of change | 9 weeks
  Assessed using the Global Perception of Change scale (answer is given using a 7-point likert scale from 1- no change to 7 - a great deal better and a considerable improvement that has made all the difference)
Perception of change | 6 months
  Assessed using the Global Perception of Change scale (answer is given using a 7-point likert scale from 1- no change to 7 - a great deal better and a considerable improvement that has made all the difference)

CONTACTS AND LOCATIONS:
Locations (1):
- School of Health Sciences, Aveiro, Portugal

REFERENCES:
- [Derived] Heleno E, Andias R, Neto M, Silva AG. A Feasibility Study of Pain Neuroscience Education and Exercise for Community-Dwelling Older Adults With Chronic Pain. J Geriatr Phys Ther. 2023 Jan-Mar 01;46(1):26-35. doi: 10.1519/JPT.0000000000000327. Epub 2021 Aug 19. PMID 34417415